CLINICAL TRIAL: NCT06179446
Title: A PHASE 1, RANDOMIZED, OBSERVER-BLIND, DOSE-RANGING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MODIFIED RNA VACCINE CANDIDATES AGAINST PANDEMIC INFLUENZA IN HEALTHY ADULTS
Brief Title: A Study to Learn How Safe, Tolerable and Capable of Producing an Immune Response is, a Modified RNA Vaccine Against Pandemic Influenza
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C5561001; NCT06179446 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Grippe; Influenza; Vaccines
Keywords: Flu; Pandemic influenza; RNA vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- pdmFlu vaccine 1 (Experimental)
  Interventions: Biological: pdmFlu vaccine
- pdmFlu vaccine 2 (Experimental)
  Interventions: Biological: pdmFlu vaccine
- pdmFlu vaccine 3 (Experimental)
  Interventions: Biological: pdmFlu vaccine
- pdmFlu vaccine 4 (Experimental)
  Interventions: Biological: pdmFlu vaccine
- pdmFlu vaccine 5 (Experimental)
  Interventions: Biological: pdmFlu vaccine
- pdmFlu vaccine 6 (Experimental)
  Interventions: Biological: pdmFlu vaccine
- pdmFlu vaccine 7 (Experimental)
  Interventions: Biological: pdmFlu vaccine
- pdmFlu vaccine 8 (Experimental)
  Interventions: Biological: pdmFlu vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Licensed influenza vaccine (Active Comparator)
  Interventions: Biological: Licensed influenza vaccine

INTERVENTIONS:
Biological: pdmFlu vaccine — Intramuscular injection
  Arms: pdmFlu vaccine 1; pdmFlu vaccine 2; pdmFlu vaccine 3; pdmFlu vaccine 4; pdmFlu vaccine 5; pdmFlu vaccine 6; pdmFlu vaccine 7; pdmFlu vaccine 8
Biological: Placebo — Intramuscular injection
  Arms: Placebo
Biological: Licensed influenza vaccine — Intramuscular injection
  Arms: Licensed influenza vaccine

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study vaccine for the possible prevention of influenza. Influenza is a disease that can spread easily from one person to another and cause body aches, fever, cough, and other symptoms. The study vaccine is called Pandemic Influenza modRNA (pdmFlu) Vaccine.

This study is seeking for participants who are:

* between the ages of 18 to 49 years old or 65 to 84 years old.
* willing and able to follow with all scheduled visits, treatment plan, laboratory tests, lifestyle changes, and other study procedures.
* healthy as confirmed by medical history, physical examinations, and the study doctor.
* capable of signing informed consent.

Participants will receive either:

* the pdmFlu vaccine,
* a licensed influenza vaccine
* a placebo. A placebo does not have any medicine in it but looks just like the study medicine.

Participants will not know which vaccine they receive. Participants will receive the study vaccines as a single shot in the arm. The study will compare participant experiences to help understand if the pdmFlu vaccine is safe and effective. Participants will take part in this study for up to 13 months. During this time, the participants will receive the study vaccine and take part in follow-up visits.

ELIGIBILITY:
Key Inclusion Criteria:

- Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Key Exclusion Criteria:

- Does not meet seasonal influenza vaccine requirements per cohort.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Percentage of participants by age group reporting local reactions | For 7 days after vaccination
Percentage of participants by age group reporting systemic events | For 7 days after vaccination
Percentage of participants by age group reporting adverse events | From vaccination to 4 weeks after each vaccination
Percentage of participants by age group reporting serious adverse events | From vaccination to 6 months after last vaccination or through the last visit, whichever is longer
Percentage of participants by age group reporting medically attended adverse events | From vaccination to 6 months after last vaccination or through the last visit, whichever is longer
Percentage of participants by age group with abnormal hematology and chemistry laboratory values | 1 week, 3 weeks, 6 weeks, 8 weeks and 12 weeks after vaccination 1, 1 week and 4 weeks after vaccination 2, 1 week and 4 weeks after booster vaccination
Percentage of participants by age group with grading shifts in hematology and chemistry laboratory assessments | Between baseline and 1 week, 3 weeks, 6 weeks, 8 weeks and 12 weeks after vaccination 1, 1 week and 4 weeks after vaccination 2, 1 week and 4 weeks after booster vaccination
Percentage of participants by age group with new clinically significant ECG abnormalities | 1 week, 3 weeks, 6 weeks, 8 weeks and 12 weeks after vaccination 1, 1 week and 4 weeks after vaccination 2, 1 week and 4 weeks after booster vaccination
Percentage of participants by age group with new troponin I abnormalities | 1 week, 3 weeks, 6 weeks, 8 weeks and 12 weeks after vaccination 1, 1 week and 4 weeks after vaccination 2, 1 week and 4 weeks after booster vaccination

SECONDARY OUTCOMES:
Geometric mean titers (GMTs) of hemagglutination inhibition (HAI) titers | At baseline, 1 week, 3 weeks, 6 weeks, 8 weeks and 12 weeks, 16 weeks and 6 months after vaccination 1, 1 week, 4 weeks, 3 months and 6 months after vaccination 2, 1 week, 4 weeks, 12 weeks and 6 months after booster vaccination
Geometric mean fold rise (GMFR) in HAI titers from before vaccination to each subsequent timepoint | At baseline, 1 week, 3 weeks, 6 weeks, 8 weeks and 12 weeks, 16 weeks and 6 months after vaccination 1, 1 week, 4 weeks, 3 months and 6 months after vaccination 2, 1 week, 4 weeks, 12 weeks and 6 months after booster vaccination
Proportion of participants by age group achieving HAI seroconversion | At baseline, 1 week, 3 weeks, 6 weeks, 8 weeks and 12 weeks, 16 weeks and 6 months after vaccination 1, 1 week, 4 weeks, 3 months and 6 months after vaccination 2, 1 week, 4 weeks, 12 weeks and 6 months after booster vaccination
Proportion of participants by age group with HAI titer >=1:40 | At baseline, 1 week, 3 weeks, 6 weeks, 8 weeks and 12 weeks, 16 weeks and 6 months after vaccination 1, 1 week, 4 weeks, 3 months and 6 months after vaccination 2, 1 week, 4 weeks, 12 weeks and 6 months after booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut
  - Research Centers of America, Hollywood, Florida
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5561001